CLINICAL TRIAL: NCT00923780
Title: Prospective Evaluation of Tumor Angiogenesis in Endocrine Neoplasms
Brief Title: Evaluation of Blood Vessel Formation in Endocrine Tumors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070060; 07-C-0060; NCT00898729 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-28

CONDITIONS: Lesions
Keywords: Tissue Acquisition; Gene Expression; Class Predictor Model; Endocrine Tumor
MeSH Terms: conditions — Endocrine Gland Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Tumors depend on blood vessels to provide the nourishment that allows them to grow.
* Thyroid, parathyroid, adrenal gland and pancreatic neuroendocrine tumors are among the tumors that contain the most blood vessels. Thus, endocrine tumors are important for the study of new blood vessel formation in tumors.

Objectives:

-To obtain tissues from endocrine tumors for examination to determine how they differ from normal tissue.

Eligibility:

-Patients who are scheduled for surgery to remove an endocrine tumor, those in or around the thyroid, parathyroid, adrenal gland, pancreas, or any neuroendocrine tissue.

Design:

* Tissues will be obtained from patients during surgery to remove thyroid, parathyroid, adrenal, pancreas, or neuroendocrine tumors.
* About 400 patients will be enrolled in the study over a period of 5 years.

DETAILED DESCRIPTION:
Background:

* Endocrine neoplasms are among the fastest growing tumors in incidence in the United States. Between 1995 and 2005, the incidence of thyroid carcinoma has increased 98 percent.
* Tumors of the thyroid, parathyroid, adrenal gland and pancreatic neuroendocrine tumors are among some of the most highly vascularized tumors seen.
* Consequently, endocrine neoplasms provide an extremely important model for the study of tumor angiogenesis.
* The Tumor Angiogenesis Section of the Surgery Branch, NCI has a focus on studying neovascular formation in neoplastic tissues. In addition, this section has primary responsibility for providing endocrine surgery consultative services to the NIH. As such, our Section is uniquely positioned to acquire and perform important studies on endocrine tissue to help advance our knowledge of the mechanisms involved in tumor vessel development. The majority of the patients enrolled on this study will be patients on other protocols throughout the NIH, for which our Section is consulted in order to perform their surgery.

Objectives:

Primary Objective:

-To develop a class predictor model based on gene expression patterns to distinguish benign from neoplastic endocrine tissue for each of the endocrine histologies under study. This objective will drive the statistical endpoints of the study.

Secondary Objectives:

* To utilize the tissue obtained from these endocrine neoplasms for studies of gene expression changes, proteomic changes, and methylation changes.
* To perform histologic examination of these tissues including immunohistochemistry and in situ hybridization in order to study changes in tumor neovessel formation.
* To obtain, when accessible, adjacent normal endocrine tissue for comparison with the neoplastic tissue.
* To collect tissues from endocrine neoplasms arising in the thyroid, parathyroid, adrenal, pancreas, and extraadrenal neuroendocrine rests for future analysis and correlation with clinical outcome.

Eligibility:

* Patients with radiographic evidence of, biochemical evidence of, or histologically/cytologically proven, endocrine neoplasms, including lesions of the thyroid, parathyroid, adrenal, extra-adrenal endocrine rests, paragangliomas, neuroblastomas and pancreas.
* Patients must have an ECOG performance score of 0-2.
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery.

Design:

* A tissue acquisition trial in which tissues will be obtained at the time of surgical operation for the removal of neoplasms of the thyroid, parathyroid, adrenal, pancreas, paragangliomas and or extraadrenal rests of neuroendocrine tissue.
* Tissue will be processed at the time of collection, stored and then shipped to the PI's laboratory for further processing.
* No investigational therapy will be given.
* It is anticipated that 400 patients will be enrolled over a period of 5 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients referred to the Endocrine Consult Service with radiographic evidence of, biochemical evidence of, or histologically/cytologically proven, endocrine neoplasms, including lesions of the thyroid, parathyroid, adrenal, extra-adrenal endocrine rests, paragangliomas, neuroblastomas and pancreas.
* Patients must have an ECOG performance score of 0-2.
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery.
* Patients undergoing treatment for their neoplasm may be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2007-01-05; Primary Completion 2009-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mazzanti C, Zeiger MA, Costouros NG, Umbricht C, Westra WH, Smith D, Somervell H, Bevilacqua G, Alexander HR, Libutti SK. Using gene expression profiling to differentiate benign versus malignant thyroid tumors. Cancer Res. 2004 Apr 15;64(8):2898-903. doi: 10.1158/0008-5472.can-03-3811. PMID 15087409
- [Background] Libutti SK, Crabtree JS, Lorang D, Burns AL, Mazzanti C, Hewitt SM, O'Connor S, Ward JM, Emmert-Buck MR, Remaley A, Miller M, Turner E, Alexander HR, Arnold A, Marx SJ, Collins FS, Spiegel AM. Parathyroid gland-specific deletion of the mouse Men1 gene results in parathyroid neoplasia and hypercalcemic hyperparathyroidism. Cancer Res. 2003 Nov 15;63(22):8022-8. PMID 14633735
- [Background] Bergers G, Javaherian K, Lo KM, Folkman J, Hanahan D. Effects of angiogenesis inhibitors on multistage carcinogenesis in mice. Science. 1999 Apr 30;284(5415):808-12. doi: 10.1126/science.284.5415.808. PMID 10221914